CLINICAL TRIAL: NCT04433390
Title: Time to Transit Recovery After Treatment With Naloxegol in Cardiac Surgery Intensive Care Trial
Brief Title: Effect of Naloxegol on Postoperative Ileus in Patients Undergoing Cardiac Surgery
Acronym: TRANSIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-09
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Ileus (Post Cardiac Surgery Constipation)
Keywords: Opioid induced constipation; cardiac surgery; transit recovery
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the nurse giving the treatment is not the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxegol group (Experimental): naloxégol tablet by oral route
  Interventions: Drug: Naloxegol
- Placebo group (Placebo Comparator): inert tablet by oral route
  Interventions: Drug: inert tablet

INTERVENTIONS:
Drug: Naloxegol — one naloxegol 12.5 mg tablet will be administrated 2 hours before surgery. One 25 mg naloxegol tablet per day will be administrated from 24h post-surgery until bowel movement; for maximum 5 days.
  Arms: Naloxegol group
Drug: inert tablet — one inert tablet will be administrated 2 hours before surgery. One inert tablet per day will be administrated from 24h post-surgery until bowel movement; for maximum 5 days.
  Arms: Placebo group

SUMMARY:
Postoperative ileus, defined as the transient postoperative functional inhibition of propulsive bowel activity, commonly occurs in patients after cardiac surgery and contributes to postoperative morbidity.

Naloxegol is a peripheral opioid receptor antagonist. Recent studies showed that naloxegol is effective in the treatment of chronic opioid-induced constipation but there is no data on its use in the management of postoperative ileus after cardiac surgery.

The main objective of this prospective, double-blind, randomized, placebo-controlled trial is to assess the effectiveness of the perioperative use of naloxegol in reducing the duration of the postoperative ileus in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Digestive complications following cardiac surgery, such as paralytic ileus and Ogilvie syndrome, are frequent and worsen the prognosis of patients. They pose a real problem of care in intensive care, inducing morbidity and mortality, extended hospital stay and a significant post-operative cost.

Few treatments are effective to reduce transit recovery time, except the neostigmine which has a serious side effects including cardiac ones.

During cardiac surgery, opioid treatments are frequently used to relieve the pain like sternotomy pain.

The pharmacologic effect of opioid induces the postoperative uleus. Opioid receptors are distributed in the central nervous system, where they are involved in the perception of pain, and in the peripheral nervous system, especially in the mesenteric nervous system, where they regulate intestinal peristalsis.

Morphine receptors antagonist are a target for prevention and treatment of post operative ileus syndrome such as alvimopan and naloxone.

A therapeutic trial demonstrates a decrease in the rate of pneumonia in intensive care patient mechanically ventilated who received naloxone.

Naloxegol is a peripheral antagonist of opioid receptor, from the alvimopan family. It has been designed to antagonize the peripheral, but not central, effects of opioids at therapeutic doses. Naloxegol is a substrate for cytochrome P450 (CYP 3A4). Following oral administration, naloxegol is absorbed rapidly, with peak concentrations achieved at less than 2 hours.

After once daily administration, plasma concentration equilibrium is reached within 2-3 days with minimal accumulation.

The main route of elimination for naloxegol is hepatic. Naloxegol has been shown to be effective in randomized trials of chronic opioid induced constipation, but there is no data on its use in the postoperative ileus.

Research hypothesis: the addition of naloxegol in pre and postoperative cardiac surgery could reduce the time to transit recovery and the rate of digestive and respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old,
* Undergoing cardiac surgery with cardiopulmonary bypass,
* For women of child bearing potential without contraception, beta-HCG negative result
* Having signed a written informed consent form,
* Affiliation to the social security system.

Exclusion Criteria:

* Allergy or known hypersensitivity to Naloxegol or any of the excipients or any other opioid antagonist
* Pregnant or breastfeeding women
* Severe hepatic failure, history of cirrhosis
* Moderate or severe renal failure (GFR<60ml/min)
* Concomitant treatment with a strong cytochrome P450 3A4 inhibitor
* History of acute gastro-intestinal obstruction known or suspected
* History of digestive arteritis
* Clinically relevant alteration of the blood-brain-barrier
* Cancer with increased risk of gastro-duodenal perforation
* Disorder that could alter the integrity of the gastrointestinal lining
* Regular treatment with laxative drugs
* Concomitant treatment with methadone
* Patient unable to take a drug by oral route
* Patient under protection of the adults (guardianship, curators or safeguard of justice),
* Patient included or planning to be included in another research protocol relating to medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of perioperative naloxegol administration on the duration of postoperative ileus after cardiac surgery | 5 days
  Time (hour) to transit recovery after cardiac surgery

SECONDARY OUTCOMES:
Incidence of digestive complications | 30 days
  rate of digestive complications
Evaluate the effect of the administration of Naloxegol on respiratory complications | 30 days
  rate of respiratory complications
Evaluate the effect of the administration of Naloxegol on infectious complications | 30 days
  rate of infectious complications
Verify the effectiveness of analgesia | day 1, day2, day3
  Pain Visual Analogue Scale (VAS) ranging from 0 to 10 (0=no pain, 10=worst possible pain)
Compare the length of hospital stay | 30 days
  Duration of hospital stay (days)
Compare the length of ICU stay | 30 days
  Duration of ICU stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Neuilly Sur Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laghlam D, Gibert H, Merzoug M, Leclerc D, Coroyer L, Estagnasie P, Squara P, Nguyen LS, Geri G. Effects of naloxegol on transit recovery in patients undergoing cardiac surgery: A randomized, double-blind, placebo-controlled trial. Anaesth Crit Care Pain Med. 2025 Apr;44(2):101498. doi: 10.1016/j.accpm.2025.101498. Epub 2025 Feb 21. PMID 39988233